CLINICAL TRIAL: NCT00323908
Title: QM-MSP, Ki-67, and Cytomorphology of RPFNA Specimens From High Risk Women
Brief Title: Protocol to Examine Methylation of Tumor Suppression Genes in Women at High Risk of Developing Breast Cancer
Status: Completed | Type: Observational
Sponsor: Carol Fabian, MD (Other)
Collaborators: University of Alabama at Birmingham (Other); Avon Foundation (Other); National Cancer Institute (NCI) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 9933
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; prevention; tissue sampling; polymorphisms; steroid and carcinogen metabolism
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women at high risk for developing breast cancer

SUMMARY:
A study to examine the correlations between methylation of various genes associated with breast cancer and proliferation and cytomorphology in breast epithelial cells acquired by random periareolar fine needle aspiration of women at high risk for development of breast cancer.

DETAILED DESCRIPTION:
A study to examine the correlation between gene promotor methylation and benign breast tissue proliferation and cytomorphology collected via random periareolar fine needle aspiration in postmenopausal women at increased risk for breast cancer.

ELIGIBILITY:
Inclusion criteria:

* women at high risk of developing breast cancer determined by family or personal history
* willing to participate in companion protocol (KUMC HSC#4601) for random periareolar fine needle aspiration (RPFNA) for correlational studies

Exclusion criteria:

* exclude women who have been on raloxifene, tamoxifen, letrozole, anastrozole or exemestane within the six months prior to RPFNA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical center
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2005-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center